CLINICAL TRIAL: NCT04370769
Title: Understanding Perception of Risk in Pregnancy Associated Progression of Chronic Kidney Disease
Brief Title: PREDICT: Thinking About Pregnancy Risk in Women With Kidney Disease
Acronym: PREDICT_RP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT_RP
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Diseases; Pregnancy Related
Keywords: Risk perception
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Kidney Disease: Women with kidney disease

SUMMARY:
Currently, there is no robust evidence about how women with Chronic Kidney Disease (CKD) perceive pregnancy risk. The aims of this research are to understand women with CKD's perception of risk in pregnancy. In order to provide appropriate pre-pregnancy and antenatal counselling including accurate presentation of risk of pregnancy outcomes, it is important to establish how do women with CKD perceive their risk in pregnancy. In addition, to facilitate discussion about pregnancy for women with CKD, it is critical to understand key psychosocial factors influencing their risk perceptions.

This study will be conducted in two phases. In phase one, risk perceptions in women with CKD who are contemplating pregnancy will be quantitatively measured with potential influencing psychosocial factors including their illness perceptions, quality of life, anxiety, depression and perceived social support. Demographic, pregnancy-intentions, medical and pregnancy histories will also be collected. Phase one findings will establish to what extent do women with CKD perceive their pregnancy risk.

In phase two, perception of risk, pregnancy intention and behaviour, will be qualitatively explored in women with CKD who perceive high and low degrees of risk. This sub-study will facilitate understanding about which factors and experiences impact risk perception and their relationship with pregnancy intentions and behaviour.

DETAILED DESCRIPTION:
The objectives for this research are:

1. To understand how women with CKD perceive their pregnancy risk.
2. To examine the associations between biopsychosocial factors (demographics, psychosocial factors, renal and pregnancy history) and women with CKD's perception of risk in pregnancy.
3. To examine the relationship between pregnancy-related intention and perception of pregnancy risk in women with CKD.
4. To gain an in-depth understanding of the biopsychosocial factors which influence risk perception and pregnancy-related behaviour, in women with CKD who perceive high and low risk perceptions.

To achieve these objectives this study is divided into two phases:

Phase 1: Quantitative assessment of risk perception and biopsychosocial factors in women with CKD Phase 2: Qualitative exploration of risk perception in women with CKD with high and low risk perception scores

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CKD stages 1-5 according to KDOQI guidelines)

  * ≥18 years old
  * Planning a pregnancy
  * Adults who have the capacity/capability to provide fully informed consent for the study

Exclusion Criteria:

* Already established on haemodialysis or peritoneal dialysis
* Women < 18 years old or >50 years old
* Inability or unwilling to give informed consent
* Does not speak English

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with CKD who are planning a pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Pregnancy intention | Baseline (Pre-pregnancy)
  Measuring women's pregnancy intention using standardised measure (Desire to Avoid Pregnancy Questionnaire)
Risk perception of pregnancy risk (Perception of Pregnancy Risk Questionnaire) | Baseline (Pre-pregnancy)
  Measuring women's perception of pregnancy risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Elizabeth Ralston, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ralston ER, Smith P, Clark K, Wiles K; RaDaR CKD Pregnancy Group; Chilcot J, Bramham K. Exploring biopsychosocial correlates of pregnancy risk and pregnancy intention in women with chronic kidney disease. J Nephrol. 2023 Jun;36(5):1361-1372. doi: 10.1007/s40620-023-01610-2. Epub 2023 Mar 27. PMID 36971978